CLINICAL TRIAL: NCT02455037
Title: Evaluation of a Neck Strengthening Program as a Potential Intervention to Reduce the Risk of Sport-related Concussion
Brief Title: Evaluation of a Neck Strengthening Program to Reduce the Risk of Sport-related Concussion
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Michigan (Other)
Responsible Party: Principal Investigator, James Eckner, Assistant Professor, University of Michigan
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: HUM00087641
Record Dates: First submitted 2015-05-14; First posted 2015-05-27 (Estimated); Last update posted 2021-08-31 (Actual); Status verified 2021-08

CONDITIONS: Sport-related Concussion; Brain Concussion; Healthy
Keywords: Concussion; Contact sport; Collision sport; Neck strengthening
MeSH Terms: conditions — Brain Concussion

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Body Strengthening (Only) (No Intervention): All participants will complete a general resistance exercise training program.
- Body Strengthening + Neck Strengthening (Experimental): Participants assigned to the neck strengthening group will complete additional supervised exercises specifically designed to strengthen the neck.
  Interventions: Other: Neck Strengthening

INTERVENTIONS:
Other: Neck Strengthening — Targeted neck strengthening exercises
  Arms: Body Strengthening + Neck Strengthening

SUMMARY:
Evaluation of a neck strengthening program as a potential intervention to reduce the risk of sport-related concussion in youth contact and collision sport athletes.

DETAILED DESCRIPTION:
This is a pilot study to investigate the effect of a supervised 8 week strengthening intervention in male and female youth contact and collision sport athletes. Participants will complete a supervised strengthening exercise intervention involving manual resistance exercises administered by a strength coach with pre- and post-intervention assessments of neck size and strength.

ELIGIBILITY:
Inclusion Criteria:

* Contact/collision sport athletes (for example, american football, soccer, rugby, lacrosse, ice hockey, field hockey, basketball, wrestling, boxing, martial arts, water polo)

Exclusion Criteria:

* History of concussion (suspected or diagnosed) in the previous 6 months
* History of neck pain or injury in the previous 6 months
* History of migraine headaches
* History of personal or parental history of a diagnosed anxiety disorder

Ages: 12 Years to 19 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 17 (Actual)
Dates: Start 2015-05; Primary Completion 2015-10 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Head linear velocity | Change from baseline to end of 8 week intervention.
Head angular velocity | Change from baseline to end of 8 week intervention.

OTHER OUTCOMES:
Neck size (girth and muscle cross-sectional area) | Change from baseline to end of 8 week intervention.
Neck strength (maximum force generating capacity) | Change from baseline to end of 8 week intervention.

CONTACTS AND LOCATIONS:
Overall Officials: James T Eckner, MD, MS, Principal Investigator — Assistant Professor, Department of Physical Medicine & Rehabilitation
Locations (1):
- University of Michigan, Ann Arbor, Michigan, United States

REFERENCES:
- [Background] Ashton-Miller JA, McGlashen KM, Herzenberg JE, Stohler CS. Cervical muscle myoelectric response to acute experimental sternocleidomastoid pain. Spine (Phila Pa 1976). 1990 Oct;15(10):1006-12. doi: 10.1097/00007632-199015100-00005. PMID 2263964
- [Background] Centers for Disease Control and Prevention (CDC). Nonfatal traumatic brain injuries from sports and recreation activities--United States, 2001-2005. MMWR Morb Mortal Wkly Rep. 2007 Jul 27;56(29):733-7. PMID 17657206
- [Background] Dvir Z, Prushansky T. Cervical muscles strength testing: methods and clinical implications. J Manipulative Physiol Ther. 2008 Sep;31(7):518-24. doi: 10.1016/j.jmpt.2008.08.008. PMID 18804002
- [Background] Eckner JT, Oh YK, Joshi MS, Richardson JK, Ashton-Miller JA. Effect of neck muscle strength and anticipatory cervical muscle activation on the kinematic response of the head to impulsive loads. Am J Sports Med. 2014 Mar;42(3):566-76. doi: 10.1177/0363546513517869. Epub 2014 Jan 31. PMID 24488820
- [Background] Broglio SP, Sosnoff JJ, Shin S, He X, Alcaraz C, Zimmerman J. Head impacts during high school football: a biomechanical assessment. J Athl Train. 2009 Jul-Aug;44(4):342-9. doi: 10.4085/1062-6050-44.4.342. PMID 19593415
- [Background] Dick RW. Is there a gender difference in concussion incidence and outcomes? Br J Sports Med. 2009 May;43 Suppl 1:i46-50. doi: 10.1136/bjsm.2009.058172. PMID 19433425
- [Background] Garces GL, Medina D, Milutinovic L, Garavote P, Guerado E. Normative database of isometric cervical strength in a healthy population. Med Sci Sports Exerc. 2002 Mar;34(3):464-70. doi: 10.1097/00005768-200203000-00013. PMID 11880811
- [Background] Guskiewicz KM, Mihalik JP. Biomechanics of sport concussion: quest for the elusive injury threshold. Exerc Sport Sci Rev. 2011 Jan;39(1):4-11. doi: 10.1097/JES.0b013e318201f53e. PMID 21088602
- [Background] Hamilton DF, Gatherer D, Jenkins PJ, Maclean JG, Hutchison JD, Nutton RW, Simpson AH. Age-related differences in the neck strength of adolescent rugby players: A cross-sectional cohort study of Scottish schoolchildren. Bone Joint Res. 2012 Jul 1;1(7):152-7. doi: 10.1302/2046-3758.17.2000079. Print 2012 Jul. PMID 23610685